CLINICAL TRIAL: NCT06830330
Title: Effect of Virtual Reality Application on Anxiety and Fear in Patients Undergoing Laparoscopic Abdominal Surgery: A Randomized Controlled Study
Brief Title: Effect of Virtual Reality Application on Anxiety and Fear in Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Nursevim Aydıngülü, Research assisstant, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sağlık Bilimleri Fakültesi
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Preoperative Patients; Patients Undergoing Abdominal Surgery
Keywords: preoperative anxiety; surgical fear; virtual reality; Anxiety State
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study was conducted as a randomized, controlled, interventional study.
Who Masked: Participant
Masking Description: Participants were blinded using a single-blind method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Group (Experimental): Virtual Reality Group
  Interventions: Behavioral: Virtual reality
- Control Group (No Intervention): Control group

INTERVENTIONS:
Behavioral: Virtual reality — Patients in the experimental group were shown videos of natural landscapes with VR glasses in their beds. This application was used to distract patients who were experiencing negative emotions just before surgery. The video session begins with the introduction of the virtual reality glasses. A motionless virtual area is determined at the point where the patient's stretcher is located. The glasses are placed on the patient's head and both hands of the patient are trained to use the remote control. Video content is selected and started according to the patient's preference. Video sessions last approximately 10 minutes.
  Arms: Virtual Reality Group

SUMMARY:
The goal of this clinical trial is to learn if virtual reality application effects on anxiety and fear in patients who will undergo abdominal surgery.

It will also learn about the practical of virtual reality application in preoperative theatre. The main questions it aims to answer are:

* Does virtual reality reduce patient anxiety levels before surgery?
* Is virtual reality useful for patients to watch videos in the preoperative area? Researchers will compare virtual reality videos to routine nursing care to see if virtual reality works to treat preoperative anxiety and surgical fear.

Participants will:

* watch videos of nature scenes with VR glasses in the waiting area before surgery.
* answer the surgical fear quastionairre items for preoperative fear test

DETAILED DESCRIPTION:
Research Design This study aims to determine the effect of virtual reality glasses on the anxiety and fear experienced by patients undergoing abdominal surgery. The randomized, controlled and interventional study blinded the participants using a single-blind method.

Participants The study was conducted in the general surgery clinic of Balcalı Hospital Health Application and Research Center and the waiting room (preoperative area) of the operating room affiliated to this clinic. The research universe consisted of patients who were examined in the general surgery clinic and planned to undergo abdominal surgery under general anesthesia using the laparoscopic method. For this purpose, the researchers conducted a preliminary interview with the patients admitted to the clinic the night before the surgery. Among the patients who were interviewed, patients who were able to communicate and accepted to participate in the study, aged over 18 were included. Patients who used glasses, had an ASA score above 3, had vertigo and motion sickness-motion sickness, and had a known psychiatric or behavioral diagnosis were excluded from the study.

The study was based on the study by Gökçe and Arslan (2023), and when type 1 error was taken as 0.05, power was taken as 80%, and effect size was taken as 0.86, the sample size was calculated as 46 in total, 23 in both groups, in order to find a significant difference between the groups. The included patients were divided into intervention and control groups with simple randomization method. The study was completed by analyzing the data of 24 patients in the experimental group and 23 patients in the control group.

Data Collection During the data collection phase, the "Patient Introduction Form" created in line with the literature was used to define the sociodemographic characteristics of the participants. For other parameters; "State-Trait Anxiety Inventory", "Surgical Fear Scale" were used.

Patient Introduction Form: The section containing the patient's demographic data includes questions regarding age, gender, body mass index, education, marital status, presence of chronic disease, surgical experience, smoking, preoperative fasting period and the type of surgery to be performed.

Surgical Fear Scale: It was developed by Theunissen and colleagues in 2014 to determine the level of fear experienced by patients scheduled for surgical treatment due to short- and long-term outcomes of the surgical procedure. The Turkish validity and reliability of the scale was performed by Bağdigen and Karamanözlü in 2018. The scale, consisting of 8 items, is scored between 0 and 10. A score of 0 for each item means "I am not afraid at all", while a score of 10 means "I am very afraid". The scale consists of two sub-dimensions regarding the source of fear. The first 4 items of the scale measure the fear of short-term outcomes of surgery, while the last 4 items measure the fear of long-term outcomes. The lowest score that can be obtained from the sub-dimensions in the scale is 0, and the highest score is 40. The sum of the two sub-dimension scores gives the total score of the scale. The lowest total score of the scale is 0, and the highest total score is 80. A high score indicates that the fear of surgery is high.

State and Trait Anxiety Inventory (STAI-I): The state anxiety scale shows how individuals feel at a certain moment and under a certain condition, while the trait anxiety scale shows how they feel in general. The scale was developed by Spielberger in 1970. The scale, which was adapted to Turkish by Öner and Le Compte in 1983, consists of a total of 40 items. The first 20 items of the scale examine the individual's state anxiety, and the last 20 items examine the individual's trait anxiety, totaling 40 items. Each item is scored on a 4-point Likert type. In the state anxiety scale, 1 point means "not at all", 2 means "a little", 3 means "a lot of the time", and 4 points means "completely". Scores in the trait anxiety scale are as follows; 1 means "almost never", 2 means "sometimes", 3 means "a lot of the time", 4 means "almost always". A total score of 20-80 can be obtained from both scales. A high score indicates a high level of anxiety. Two separate keys are prepared to determine the total weights of direct and reversed expressions. The total weighted score of the reversed expressions is subtracted from the total weight score of the direct expressions. A previously determined and unchanging value is added to the number found. This unchanging value is 50 for state anxiety and 35 for trait anxiety. The resulting value shows the individual's anxiety score. The total score obtained from both scales varies between 20 and 80. A high score indicates a high level of anxiety, while a low score indicates a low level of anxiety.

2.723 / 5.000 Data Collection Process During the data collection process, the researchers met with patients who met the inclusion criteria in the clinic the night before the surgery and obtained written consent to participate in the study. A total of 84 patients were evaluated for research eligibility. Of these patients, 23 were excluded from the study because they did not meet the inclusion criteria, and 5 were excluded because they did not accept participation. During the preliminary interview (Time 1), written consent to participate in the study was obtained from patients who met the inclusion criteria. Patients who accepted participation were administered the patient identification form and trait anxiety scale. They were also informed that they would be interviewed again the next morning before surgery. Patients who accepted participation were assigned to one of the study groups according to the determined randomization method on the morning of the surgery (Time 2). Randomization of the patients was performed according to the study days. Data from the experimental group were collected on three days of the week, and data from the control group were collected on two days. During the data collection process, the days determined for the experimental group and the control group were randomized each week. Thus, patients were blinded in terms of the applications in the study groups. The patient identification form, trait anxiety scale, state anxiety scale and surgical fear scale were first administered to patients in the preoperative waiting unit.

Then, the patients in the experimental group were shown videos containing natural scenes with the help of VR glasses (Oculus Quest 2, 64GB) in the patient bed. This application was used to divert the attention of patients experiencing negative emotions just before surgery. The video session begins with the introduction of the virtual reality glasses. A motionless virtual area is determined at the point where the patient's stretcher is located. The glasses are placed on the patient's head and both hands of the patient are trained to use the remote control. The video content is selected and started according to the patient's preference. The video sessions last approximately 10 minutes. Patient-specific preparation procedures (opening vascular access, taking vital signs, premedication, informing the patient, etc.) were performed for the patients in the control group. The state anxiety scale and surgical fear scale were repeated for both groups 15 minutes after the procedures determined for the application and control groups were applied (Time 3).

6 of the patients in the experimental group and 2 of the patients in the control group were excluded from the study because the posttest could not be applied when they were taken into surgery. In addition, one patient experienced dizziness and the video session was interrupted and the patient was excluded from the study. The data collection process was terminated when the number determined by power analysis was reached. The study was completed with 24 experimental and 23 control patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for abdominal surgery under general anesthesia using the laparoscopic method
* Patients who can communicate
* Patients who agree to participate in the study
* Patients over the age of 18

Exclusion Criteria:

* Patients who use glasses
* Patients with an ASA score above 3
* Patients with vertigo and motion sickness
* Patients with known psychiatric or behavioral diagnoses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
State Anxiety Level Change | The state anxiety scale were applied to the patients 15 minutes after they watched the video with virtual reality glasses.
  The effect of virtual reality intervention on preoperative anxiety level is safely evaluated.

SECONDARY OUTCOMES:
Change in fear level related to surgery | The surgical fear scale were applied to the patients 15 minutes after they watched the video with virtual reality glasses.
  The effect of virtual reality intervention on surgical fear level is safely evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Sevban A Proffessor doctor, Study Director — Çukurova University, Faculty of Health Science
Locations (1):
- Balcali Hospital Health Application and Research Center, Adana, Sarıçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Ethics committee approval was obtained for the study to be conducted. For this reason, participant data cannot be shared.

REFERENCES:
- Available data/document: ethics committee approval — https://tip.cu.edu.tr/storage/Mevzuat/Kurullar%20Y%C3%B6nergesi.pdf